CLINICAL TRIAL: NCT02537288
Title: A Phase I Single Centre, Randomized, Double Blind (Except For Moxifloxacin), Placebo And Active Controlled, Four Way Cross Over Study Investigating The Effect Of Single Therapeutic And Supra Therapeutic Doses Of Fedovapagon On The QT/QTC Interval In Healthy Volunteers Using Oral Moxifloxacin To Confirm Assay Sensitivity
Brief Title: A Study in Healthy Volunteers to Assess the Effect of Fedovapagon on the QT/QTC Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 483-012
Record Dates: First submitted 2015-08-05; First posted 2015-09-01 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: VA106483; fedovapagon; males; females; moxifloxacin; TQT; QT/QTC; ECG; Nocturia
MeSH Terms: conditions — Nocturia | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo matched to fedovapagon (Experimental): One dose of placebo (matched to fedovapagon)
  Interventions: Drug: Placebo (for fedovapagon)
- Fedovapagon 2 mg (Experimental): One dose of 2 mg fedovapagon
  Interventions: Drug: Fedovapagon
- Fedovapagon 20 mg (Experimental): One dose of 20 mg fedovapagon
  Interventions: Drug: Fedovapagon
- Moxifloxacin 400 mg (open label) (Experimental): One dose of moxifloxacin 400 mg (open label)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Fedovapagon
  Arms: Fedovapagon 2 mg; Fedovapagon 20 mg
Drug: Moxifloxacin
  Arms: Moxifloxacin 400 mg (open label)
Drug: Placebo (for fedovapagon)
  Arms: Placebo matched to fedovapagon

SUMMARY:
The purpose of this study is to assess the electrocardiogram (ECG) effects of fedovapagon dose administration relative to placebo in healthy adult male and female subjects.

DETAILED DESCRIPTION:
Regulatory guidance (ICH E14) has emphasized the need to obtain clear robust data on the effect of new chemical entities on ECG parameters with focus on cardiac repolarization as measured by the QTc duration. Though many Phase 1, 2 and 3 trials may be conducted they usually have insufficient sample size, infrequent sampling of ECG data, or the use of inadequate controls to overcome the high rate of spontaneous change in QTc duration. This has resulted in regulatory guidance recommending a dedicated or thorough trial to define the ECG effects of new drugs.

This study will be conducted in healthy volunteers to eliminate variables known to have an effect on ECG parameters (concomitant drugs, diseases, etc.). A supra-therapeutic dose of fedovapagon is required to mimic the exposure in healthy volunteers that may occur in the target population under the worst of circumstances (e.g., concomitant use of CYP3A4 inhibitor, concomitant liver disease, presence of heart disease, taking more than the clinical dose prescribed, etc.) and to allow for PK to QTc modeling to assess the effect of drug concentration on cardiac repolarization.

A cross-over trial is the preferred design as subjects act as their own controls and since there is no accumulation of any clinical relevance and the plasma concentration of parent dissipates before 24 hours, a single dose trial will be employed. During the course of the study each subject will be administered fedovapagon at both a clinical and supra-therapeutic dose, placebo and moxifloxacin (as a positive control).

The sample size is driven by the need to do a time-matched statistical analysis on the primary endpoint as per ICH E14 guidance.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent before any study-specific procedures are conducted.
* Healthy males and females 18 to 55 years of age (inclusive).
* No clinically significant abnormal physical findings.
* No clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or admission.
* Have a body mass index (BMI) ≥18.0 to ≤29.9 kg/m2 (weight: ≥50 kg and ≤100 kg) at the Screening visit.
* Be judged by the Investigator to be in good health based on medical history, physical examination, vital sign measurements and laboratory safety tests performed at the Screening visit and before the first administration of fedovapagon, moxifloxacin or placebo.
* Have no clinically significant abnormality on an ECG performed at the Screening visit and on admission to the study center.
* Have a normal resting blood pressure.
* Must be able to understand and be willing to comply with study procedures, restrictions and requirements.
* Agree to refrain from the consumption of grapefruit or grapefruit juice beginning 1 week prior to administration of the initial administration fedovapagon, moxifloxacin or placebo, throughout the trial.
* Agree to refrain from the consumption of alcohol and/or methylxanthines e.g., caffeine (coffee, tea and cola) beginning 96 hours prior to administration of the initial administration of fedovapagon, moxifloxacin or placebo, throughout the trial.
* Current non-smokers who have not used any nicotine-containing products (chewed or smoked) or replacement products including electronic cigarettes in the 45 days prior to screening.
* Woman of child-bearing potential must be using effective methods (failure rate <1%) of birth control at least 4 weeks prior to Screening until 4 weeks after the administration of fedovapagon, moxifloxacin or placebo.
* Male subjects should be willing to use a condom with spermicide during sexual activity with female partners of child-bearing potential and must not donate sperm. Female sexual partners of male subjects should be willing to avoid pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time-matched change from baseline in QTc, placebo-adjusted and corrected for heart rate | 0-48 hours

SECONDARY OUTCOMES:
Heart rate | 0-48 hours
PR interval | 0-48 hours
QRS interval | 0-48 hours
Uncorrected QT interval | 0-48 hours
ECG morphology especially on repolarization | 0-48 hours
Correlation between the QTc change from baseline and plasma concentrations of fedovapagon | 0-48 hours
Number and type of adverse events | 0-48 hours
The observed maximum plasma concentration (Cmax) | 0-48 hours
Time to reach maximum plasma concentration (tmax) | 0-48 hours
Apparent terminal half-life (t½) | 0-48 hours
Area under the plasma concentration-time curve (AUC0-t), (AUC0-24h) and (AUC0-∞) | 0-48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Georg Golor, PD Dr med, Principal Investigator — Parexel
Locations (1):
- PAREXEL Early Phase Clinical Unit Berlin, Berlin, Germany